CLINICAL TRIAL: NCT03838445
Title: RELIEVE-PAH TRIAL: REducing Right ventricuLar faIlure With thE V-waVe Shunt in Pulmonary Arterial Hypertension
Brief Title: Reducing Right Ventricular Failure in Pulmonary Arterial Hypertension (RELIEVE-PAH)
Acronym: RELIEVE-PAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: V-Wave Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL7012
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; Interatrial Shunt; Interatrial Shunting; Atrial Septostomy
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Therapy: V-Wave Shunt (Experimental): Treatment arm patients will undergo a diagnostic right heart catheterization and invasive echocardiography to determine study eligibility followed by transseptal catheterization and V-Wave Shunt implantation.
  Interventions: Device: V-Wave Interatrial Shunt

INTERVENTIONS:
Device: V-Wave Interatrial Shunt — The V-Wave Interatrial Shunt System, includes a permanent implant placed during a minimally invasive cardiac catheterization procedure using its dedicated Delivery Catheter. The device is implanted through the fossa ovals and straddles the interatrial septum.

SUMMARY:
The objectives of the RELIEVE-PAH study are to obtain first-in-human experience with the study device in patients with severe pulmonary arterial hypertension, including evidence of initial safety, device performance and possible signals of clinical effectiveness.

DETAILED DESCRIPTION:
This is a multi-national, multi-center, prospective, non-randomized, open label trial of patients implanted with the study device. A total of up to 20 patients will be implanted with the study device and followed at regular intervals for 1 year and then annually for a total of 5 years post implant.

ELIGIBILITY:
Main Inclusion Criteria:

1. Group 1 PAH (idiopathic, connective tissue disease, HIV, corrected congenital heart disease).
2. WHO Functional Class III or IV symptoms. If WHO Class III, at least 1 High-Risk characteristic or 2 Intermediate-Risk characteristics from the 2015 ESC Guidelines.
3. Receiving maximal available and tolerable pharmacological PAH therapy ≥3 months at a stable dose for ≥1 month.

Main Exclusion Criteria:

1. Resting oxygen saturation <90 % without supplemental oxygen corrected for altitude.
2. Mean Right Atrial Pressure >20 mmHg.
3. Severe restrictive or obstructive lung disease.
4. Evidence of organ dysfunction other than right heart failure.
5. Left ventricular ejection fraction <40 %.
6. Anatomical anomaly on transesophageal echocardiography or intracardiac echocardiography that precludes implantation of Shunt across fossa ovalis (FO) of the interatrial septum.
7. Inadequate vascular access for implantation of shunt, e.g. femoral venous access for transseptal catheterization and inferior vena cava (IVC) is not patent.
8. Hemodynamic heart rhythm, or respiratory instability at time of Final Exclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety-Percentage of Treatment patients experiencing major device-related adverse events | 3 months
  Percentage of Treatment group patients experiencing any device-related Major Adverse Cardiovascular or Neurological Events (MACNE) during the first 90-days after implantation
Safety-Percentage of Treatment patients experiencing any major adverse event | 3 months
  Percentage of Treatment group patients experiencing any Major Adverse Cardiovascular or Neurological Events (MACNE) during the first 90-days after implantation
Procedure Success-Percentage of patients successfully implanted with study device | 3 months
  Percentage of patients successfully implanted with the study device at the intended location across the interatrial septum during the index procedure compared to patients with attempted implantations
Device Success-Percentage of patients implanted with right to left interatrial flow | 3 months
  Percentage of patients successfully implanted with the study device with right to left interatrial flow on echocardiography at 3 months

SECONDARY OUTCOMES:
Freedom from device related MACNE at 1 and 12 months after implantation | 1 and 12 months
  Freedom from device related Major Adverse Cardiac and Neurologic Events at 1 and 12 months after implantation.
Improvement in Exercise Capacity between baseline and 12 months | 12 months
  Improvement in Exercise Capacity measured by the six minute hall walk test from baseline to 12 months
Improvement in WHO Functional Class between baseline and 12 months | 12 months
  Improvement in World Health Organization Functional Class between baseline and 12 months.
Improvement in Quality of Life between baseline and 12 months | 12 months
  Improvement in Quality of Life as measured by the SF-36 questionnaire
Improvement in Quality of Life between baseline and 12 months | 12 months
  Improvement in Quality of Life as measured by the CAMPHOR questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Victor Tapson, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (5):
- United States (3):
  - Keck Medical Center of USC, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - The Ohio State University Wexner Medical Center - Davis Heart & Lung Research Institute, Columbus, Ohio
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Canada
- Instituto Nacional de Cardiologia, Mexico City, Mexico